CLINICAL TRIAL: NCT02363283
Title: A Phase 2 Study of CDX-011 (Glembatumumab Vedotin) for Metastatic Uveal Melanoma
Brief Title: Glembatumumab Vedotin in Treating Patients With Metastatic or Locally Recurrent Uveal Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2015-00159; NCI-2015-00159 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NCI9855; 9855 (Other: University of Texas MD Anderson Cancer Center LAO); 9855 (Other: CTEP); N01CM00039 (NIH); UM1CA186712 (NIH)
Record Dates: First submitted 2015-02-13; First posted 2015-02-16 (Estimated); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Uveal Melanoma; Stage IV Uveal Melanoma AJCC v7
MeSH Terms: conditions — Uveal Melanoma | interventions — glembatumumab vedotin; CR011-vcMMAE

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (glembatumumab vedotin) (Experimental): Patients receive glembatumumab vedotin IV over 90 minutes every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Glembatumumab Vedotin; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: Glembatumumab Vedotin — Given IV
  Other Names: Antibody-Drug Conjugate CR011-vcMMAE; CDX-011; CR011-vcMMAE; CR011-vcMMAE Immunotoxin
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial studies how well glembatumumab vedotin works in treating patients with middle layer of the wall of the eye (uveal) melanoma that has spread to other parts of the body (metastatic) or has returned at or near the same place after a period of time during which the cancer could not be detected (locally recurrent). Glembatumumab vedotin may shrink the tumor by binding to tumor cells and delivering tumor-killing substances to them.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the clinical anti-tumor activity of CDX-011 (glembatumumab vedotin) as a single-agent in the treatment of patients with metastatic uveal melanoma.

SECONDARY OBJECTIVES:

I. Description of the clinical safety and benefit of CDX-011 (glembatumumab vedotin) and pharmacodynamics changes in glycoprotein NMB (glycoprotein [transmembrane] NMB) (GPNMB) expression.

TERTIARY OBJECTIVES:

I. Characterization of the anti-tumor immunophenotype of patients receiving treatment.

II. Post hoc, correlation of rash with clinical benefit, or lack of rash with lack of benefit, will also be explored.

OUTLINE:

Patients receive glembatumumab vedotin intravenously (IV) over 90 minutes every 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic or locally recurrent uveal melanoma; because histologic or cytologic confirmation of primary uveal melanoma is not always possible, confirmation of the clinical diagnosis of uveal melanoma by the treating investigator is allowed; clinical diagnosis of uveal melanoma is often made by an ophthalmologist, not by tissue diagnosis; if an ophthalmologist diagnosed and treated a patient for uveal melanoma in the past, it is sufficient for a clinical diagnosis
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded for non-nodal lesions and short axis for nodal lesions) as >= 20 mm (>= 2 cm) with conventional techniques or as >= 10 mm (>= 1 cm) with spiral computed tomography (CT) scan, magnetic resonance imaging (MRI), or calipers by clinical exam
* The study will be limited to patients who are chemotherapy naive; patients may have received prior systemic or liver-directed local therapies for advanced uveal melanoma as long as those treatments do not involve chemotherapy; this includes, but is not limited to: immunotherapy, targeted therapy, transarterial embolization, radiofrequency ablation, or cryoablation; treatment must be completed at least 28 days prior to initiation of study therapy; radiation therapy is also allowed and must be completed at least 28 days prior to initiation of study therapy; lesions treated via radiation or liver-directed therapy may not be used as target lesions unless they demonstrate growth over a minimum of 3 months on subsequent imaging
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events (CTCAE) version (V) 5 grade =< 1 (except alopecia); certain exceptions apply, such as immunotherapy-induced hypothyroidism or adrenal insufficiency or panhypopituitarism requiring stable doses of hormone replacement or rash from prior therapy
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/uL
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Total bilirubin =< 1.5 x institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal; =< 5 x institutional upper limit of normal if liver metastasis present
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 4 months after last CDX-011 (glembatumumab vedotin) dose; women of child-bearing potential must have a negative serum pregnancy test within 14 days prior to start of protocol treatment; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men and women treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of glembatumumab vedotin administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with a history of another malignancy except for those who have been disease-free for 2 years; patients with a history of definitively treated non-melanoma skin cancer or squamous cell carcinoma of the cervix are eligible; patients with definitively treated in-situ cancers are eligible, regardless of timeframe
* Patients with neuropathy > grade 1
* Patients who are receiving any other investigational agents; if the patient received a previous investigational or other agent or treatment, a washout period of 4 weeks is required
* Patients receiving any medications or substances that are substrates of cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) will be closely monitored for toxicity; as part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Human immunodeficiency virus (HIV)-positive patients on antiretroviral medications that are CYP3A4 substrates will be closely monitored; HIV-positive patients will be excluded if they have a cluster of differentiation 4 (CD4) count < 200
* Pregnant or nursing women
* Patients who have previously received CDX-011 (glembatumumab vedotin) or other monomethyl auristatin E (MMAE)-containing agents
* Patients with a history of allergic reactions attributed to compounds of similar composition to dolastatin or auristatin (e.g. Auristatin PHE, Auristatin PE, and symplostatin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sapna Patel, Principal Investigator — University of Texas MD Anderson Cancer Center LAO
Locations (25):
- United States (25):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - University of Colorado Hospital, Aurora, Colorado
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Roswell Park Cancer Institute, Buffalo, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - M D Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: October 2015 to January 2018
Pre-assignment Details: 2 participants withdrew consents prior to starting therapy and 1 failed eligibility criteria.
Period: Overall Study
Arm/Group | Treatment (Glembatumumab Vedotin)
Started | 37
Completed | 35
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Not eligible due to transaminitis | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 62 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 34
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Using Response Evaluation Criteria in Solid Tumors Version 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (PD); PD, 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Complete Response (CR), Disappearance of all target lesions
Time Frame: From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years and 10 months
Population: participants who entered study and received treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 35
Participants
  Partial Response | 2
  Stable Disease | 18
  Disease Progression | 14
  Unknown | 1

2. Secondary Outcome: The Number of Participants With Change in Glycoprotein NMB Expression on Tumor Tissue Via Immunohistochemistry
Description: Target protein expression change from baseline to after 1 cycle of treatment.
Time Frame: Baseline to up to 21 days
Population: Of 32 enrolled participants, 26 had baseline tissue available and 24 had Day 21 tissue available leaving only 22 evaluable for the secondary outcome measure: change in tumor expression from baseline to Day 21. In other words, only 22 participants had tumor collected for both baseline and Day 21 GPNMB expression.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 22
Participants | 22

3. Secondary Outcome: Progression-free Survival
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From consent to time of progression or death, whichever occurs first, assessed up to 2 years and 10 months
Population: 37 participants signed consent 1 participant withdrew consent for survival follow up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 36
months | 3.1 [1.5 to 5.6]

4. Secondary Outcome: Number of Participants With Grade 3-4 Adverse Events According to the National Cancer Institute Common Toxicity Criteria Version 4.0
Description: Toxicity will be reported by type, frequency, and severity. Only adverse events toxicity with grade 3-4 severity.
Time Frame: through 30 days post-treatment, up to 2 years and 10 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 35
Participants
  Neutropenia | 19
  Thrombocytopenia | 1
  Diarrhea | 1
  Constipation | 1
  Vomiting | 1
  Rash, maculopapular | 2
  Pruritus | 2

5. Secondary Outcome: Overall Survival
Description: Overall survival as measured from time of enrollment to time of death due to any cause.
Time Frame: From consent to time of progression or death, whichever occurs first, assessed up to 2 years and 10 months
Population: 37 participants signed consent 1 participant withdrew consent for survival follow up
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Glembatumumab Vedotin)
Number analyzed (Participants) | 36
months | 11.9 [9 to 16.9]

ADVERSE EVENTS:
Time Frame: through 30 days post-treatment, an average of 1 year
Arm/Group | Treatment (Glembatumumab Vedotin)
All-Cause Mortality (participants affected / at risk) | 1/35
Serious Adverse Events (participants affected / at risk) | 34/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Glembatumumab Vedotin) (N=35)
Neutropenia (Blood and lymphatic system disorders) | 21
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Elevated ALT/AST (Gastrointestinal disorders) | 22
Nausea (Gastrointestinal disorders) | 18
Diarrhea (Gastrointestinal disorders) | 11
Constipation (Gastrointestinal disorders) | 8
Mucositis, oral (Blood and lymphatic system disorders) | 6
Vomiting (Gastrointestinal disorders) | 5
Alopecia (Skin and subcutaneous tissue disorders) | 28
Rash, maculopapular (Skin and subcutaneous tissue disorders) | 19
Pruritus (Skin and subcutaneous tissue disorders) | 18
Leukopenia (Blood and lymphatic system disorders) | 24
Anemia (Blood and lymphatic system disorders) | 14
Lymphopenia (Blood and lymphatic system disorders) | 6
Elevated ALP (Gastrointestinal disorders) | 9
Hyperbilirubinemia (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Oral pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 20
Pain (General disorders) | 6
Chills (Gastrointestinal disorders) | 2
Flu like symptoms (General disorders) | 2
Localized edema (General disorders) | 2
Weight loss (General disorders) | 2
Peripheral Neuropathy (Nervous system disorders) | 15
Dysgeusia (Nervous system disorders) | 8
Headache (Nervous system disorders) | 3
Generalized muscle weakness (Nervous system disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Hyponatremia (Renal and urinary disorders) | 5
Hypophosphatemia (Renal and urinary disorders) | 4
Hypokalemia (Renal and urinary disorders) | 3
Hyperkalemia (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 13
Hypoalbuminemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 2
Hot flashes (Vascular disorders) | 3
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT02363283/Prot_SAP_001.pdf